CLINICAL TRIAL: NCT02234830
Title: Randomized Comparison of ExoSeal® and Angio-Seal Vascular Closure Devices: The CLOSE-UP II Trial
Acronym: CLOSE-UP II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Cordis US Corp. (Industry); Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Evald Hoej Christiansen, MD, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-68-12
Record Dates: First submitted 2014-06-06; First posted 2014-09-09 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Coronary Disease
Keywords: PCI
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exoseal closure device (Experimental): Closure device for femoral artery access closure
  Interventions: Device: Exoseal closure device
- Angio-Seal closure device (Active Comparator): Closure device for femoral artery access closure
  Interventions: Device: Angioseal closure device

INTERVENTIONS:
Device: Exoseal closure device — Closure device for femoral artery access closure
  Arms: Exoseal closure device
Device: Angioseal closure device — Closure device for femoral artery access closure
  Arms: Angio-Seal closure device

SUMMARY:
Is the ExoSeal VSD non-inferior to Angio-Seal vascular closure device (VSD) in the incidence of adverse access site related events at 30 days.

DETAILED DESCRIPTION:
Prospective, randomized (1:1) controlled, single blind, single center study in 2000 percutaneous coronary intervention (PCI) patients comparing the ExoSeal VCD (test device) to the AngioSeal VCD (standard comparator). In-hospital and 30 days safety and efficacy endpoints and 6 months safety endpoints will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Should be able to provide valid informed signed consent
* PCI procedure including treatment by balloon and/or stent
* PCI indicated by silent ischemia, stable angina pectoris, non-ST elevation myocardial infarction (NSTEMI) or ST elevation myocardial infarction (STEMI)

Exclusion Criteria:

* Only coronary angiography
* Multiple punctures
* Active infection
* Groin haematoma before the closure procedure
* Sheath size > 7 French
* Known pseudoaneurysm or arteriovenous (AV)-fistula in the ipsilateral groin
* Prior arterial surgery in abdomen and/or lower extremities
* Cardiogenic shock
* Life expectancy less than one year
* The patient is a female of childbearing potential with possible pregnancy or a positive pregnancy test within 7 days before the index procedure or is lactating
* Simultaneous or planned subsequent femoral vein access
* Allergy to any of the components in the closure material left in the groin
* Puncture on same site < 30 days
* Peripheral artery disease patients can be included at operator´s discretion except if heavy calcification is present at the access site which at the operator's discretion precludes insertion of the VCD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 818 (Actual)
Dates: Start 2012-12-21 (Actual); Primary Completion 2016-05-14 (Actual); Study Completion 2017-05-14 (Actual)

PRIMARY OUTCOMES:
Incidence at 30 days of the composite endpoint of access site related major adverse vascular events (MAVE) | 30 days
  This includes: major bleeding and/or bleeding necessitating blood transfusion, pseudoaneurysm with indication for treatment, arteriovenous fistula, groin surgery and/or possible related vascular surgery, infection needing antibiotics.

SECONDARY OUTCOMES:
Time to haemostasis from removing the sheath (AngioSeal) or inserting the device (ExoSeal) until haemostasis | participants will be followed for the duration of hospital stay, an expected average of 2 days
  Insignificant bleeding seen on the bandage or small continuous oozing is considered haemostasis. Continuous oozing will be counted as a Bleeding Academic Research Consortium (BARC) type 1 bleeding event
Device failure | 30 minutes
  Combined endpoint of any mechanic failure, deployment failure and/or immediate profuse bleeding needing prolonged manual compression. Individual endpoints will be reported.
Vasovagal reaction until 5 minutes after end of closure procedure | 30 minuts
Need for new onset of manual compression | 30 days
Pain and discomfort related to the closure procedure | Closure procedure and 30 days
  Assessed on a numerical rating scale (NRS) from 0 (no pain or discomfort) to 10 (worst possible pain or discomfort) Scripted language will be used when discussing pain scores with the patient. Pain and discomfort score will be assessed just before and immediately after the closure procedure and reported. The delta-value will be reported and compared. The patient will be given predefined standardized instructions on how to rate and that only pain and discomfort related to the closure procedure should be assessed
Time to mobilization | participants will be followed for the duration of hospital stay, an expected average of 2 days
  From start of closure procedure to patient is mobilized. Patients treated for ST-elevation myocardial infarction are assessed separately
In-hospital large groin haematoma | participants will be followed for the duration of hospital stay, an expected average of 2 days
  Larger than 5x5 cm measured by ruler in the catheterization laboratory and at discharge
Bleedings according to the BARC definitions | 30 days
  Access site related and non-access site related
Major bleeding and/or bleeding necessitating blood transfusion | 6 months
Pseudoaneurysm with indication for treatment | 30 days and 6 months
Arteriovenous fistula | 30 days and 6 months
Groin surgery and/or possible related vascular surgery | 30 days and 6 months
Infection needing antibiotics | 30 days and 6 months
Need for medical evaluation of possible closure procedure related symptom(s) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Evald H Christiansen, MD, PhD, Principal Investigator — Arhus University Hospital Skejby
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus N
  - Odense University Hospital, Odense